CLINICAL TRIAL: NCT02618824
Title: Role of Terminal Warm Blood Cardioplegia as Myocardial Protection in the Use of Histidine-Tryptophan-Ketoglutarate Cardioplegia in Complex Congenital Heart Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Pribadi W Busro, MD, MD, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01201508011
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2015-12

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Bretschneider cardioplegic solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HTK Solution (Active Comparator): Hearts will be arrested with HTK solution during cardiac operation
  Interventions: Drug: Histidine Tryptophan Ketoglutarate Solution
- HTK Solution + TWBC (Active Comparator): Hearts will be arrested with HTK solution during cardiac operation and received terminal warm blood cardioplegia before aortic cross clamp removal.
  Interventions: Drug: Histidine Tryptophan Ketoglutarate Solution; Other: Terminal Warm Blood Cardioplegia

INTERVENTIONS:
Drug: Histidine Tryptophan Ketoglutarate Solution — Hearts will be arrested with Histidine Tryptophan Ketoglutarate (HTK) solution during cardiac operation. After aortic cross clamp 50-60 ml/kg HTK will be administered
Other: Terminal Warm Blood Cardioplegia — Terminal warm blood cardioplegia (TWBC) contains 20% HTK solution and 80% blood from cardiopulmonary bypass machine. Before aortic cross clamp removal 10-15 ml/kg TWBC will be administered with temperature 34-36 oCelcius
  Other Names: Hot Shot
  Arms: HTK Solution + TWBC

SUMMARY:
Terminal warm blood cardioplegia (TWBC) has been shown to enhance myocardial protection in adult patients. Even in pediatric patients, the use of cold blood cardioplegia followed by administration of TWBC will provide cardioprotective effect similar to adult patients. Histidine-tryptophan-ketoglutarate (HTK), is attractive for cardiac surgeons because it is administered as a single dose and is claimed to offer myocardial protection for a period of up to 180 minutes allowing performance of complex procedures without interruption. Merging the use of TWBC on the use of HTK cardioplegia, especially for pediatric cardiac cases, have not been investigated. This technique is expected to provide a longer ischemic time and a protective effect against reperfusion injury.

DETAILED DESCRIPTION:
The design of this study is a randomized controlled trial in children younger than 5 years old undergoing heart surgery with cardiopulmonary bypass. The objective of this study is to assess the role of TWBC in use of HTK cardioplegia compared with the use of HTK cardioplegia alone in open heart surgery of complex congenital heart disease. This study will be conducted at the National Cardiac Centre Harapan Kita Hospital Indonesia. Surgery will be performed in the operating room of Pediatric and Congenital Cardiac Surgery Unit. This study uses non-probability consecutive sampling. The samples are all pediatric patients with complex congenital heart disease who meet the inclusion criteria and not excluded by the exclusion criteria. Patients will be divided into two groups, the treatment group who received HTK cardioplegia and TWBC, and the control group that only received HTK cardioplegia alone. Hearts will be arrested with HTK solution during cardiac operation. HTK cardioplegia will be given through the aortic root at a dose of 50-60 ml/kg after aortic cross-clamped. For the treatment group, TWBC will be given shortly before the aortic cross clamp is removed at a dose of 10 to 15 ml/kg with temperature of 34 to 36 oCelcius. TWBC is a mixture of blood and HTK kardioplegia with a composition of four to one. The outcomes of this study are malondialdehyde as a marker of reperfusion injury due to oxidative stress, caspase-3 as a marker of apoptosis, cTn-I as a marker of myocardial cell damage and the incidence of low cardiac output syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with complex cyanotic congenital heart disease who scheduled for pediatric cardiac surgery
* Aristotle score is 8 and above
* Parents of patient have written informed consent and agree to follow the research procedures

Exclusion Criteria:

* Patient diagnosed with an other congenital defect
* Patient diagnosed with rare congenital heart defect and high mortality rate (such as hypoplastic left heart syndrome)

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of Malondialdehyde levels | after induction of anaesthesia, 30 minutes and 4 hours post aortic cross clamp removal
  Malondialdehyde (MDA) is the end product of lipid peroxidation by ROS results in a state of oxidative stress, and a marker of the increase in ROS in reperfusion injury. MDA concentration in plasma of patients measured by test methods thiobarbituric acid and spectrophotometric examination.
Change of Caspase-3 levels | after induction of anaesthesia, 30 minutes post aortic cross clamp removal
  Caspase-3 is a protease, a family of cysteine proteases that act as executor in the process of apoptosis, and is used as a marker of apoptosis. The expression of caspase-3 measured quantitatively by immunohistochemistry using polyclonal antibody method cleaved caspase-3 from myocardial biopsy.
Cardiac Troponin I levels | During the first 24 hours after cross clamp removal
  Cardiac troponin I (cTnI) s a protein involved in the process of contraction of the heart, and is only found in heart cells, which will be released into the blood circulation when heart injury. CTn-I measured with Enzyme Linked Fluorescent Assay technique. Specimens for measurement of cTnI are from whole blood or serum.
Number of patients with low cardiac output syndrome | During the first 48 hours after aortic cross clamp removal
  Low cardiac output syndrome (LCOS) is a state in which clinical sign and symptoms of low cardiac output are found with or without the increasing of arterial and venous saturation gap and metabolic acidosis, the use of new inotropic, mechanical support, or other maneuvers in order to increase cardiac output. LCOS is determined by intensivist based on the clinical presentation, laboratory and inotropic scores.

SECONDARY OUTCOMES:
Inotropic Score | During the first 72 hours post cross clamp removal
  Inotropic score is a method for determining the use of inotropic drugs used by the patient. inotropic scores obtained by the following formula: Wernowsky IS = dose dopamine (mcg/kg/min) + dose dobutamine (mcg/kg/min) + 100 x doses of epinephrine (mcg/kg/min)
Postoperative Time to Extubation | up to 3 month after surgery
Postoperative Length of Stay in Intensive Care Unit | up to 3 month after surgery
Postoperative Hospital Length of Stay | up to 3 month after surgery
All cause mortality | up to 3 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pribadi W Busro, MD, Principal Investigator — National Cardiac Centre Harapan Kita Hospital
Locations (1):
- National Cardiac Centre Harapan Kita Hospital, Jakarta, Jakarta Special Capital Region, Indonesia